CLINICAL TRIAL: NCT04010435
Title: Influence of Central Versus Peripheral Vestibular Stimulation on Recovery Outcomes in Patients With Peripheral Vestibular Disorders
Brief Title: Influence of Central Versus Peripheral Vestibular Stimulation in Patients With Peripheral Vestibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Mohamed Ali Ahmed, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/002202
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Vestibular Disorders
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (r TMS group) (Active Comparator): Twenty randomly assigned patients with unilateral peripheral vestibular disorders will undergo 10 Hz rTMS to the dorsolateral prefrontal cortex of their dominant hemisphere; in addition to designed vestibular rehabilitation exercises.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Group B (Galvanic stimulation) (Active Comparator): Twenty randomly assigned patients with unilateral peripheral vestibular disorders will undergo galvanic vestibular stimulation; in addition to designed vestibular rehabilitation exercises.
  Interventions: Device: Galvanic stimulation
- Control (Group C) (No Intervention): Twenty randomly assigned patients with unilateral peripheral vestibular disorders will undergo designed vestibular rehabilitation exercises.

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — high frequency (10 HZ) rTMS pulses are applied to the dorsolateral prefrontal cortex of the dominant hemisphere.
  Arms: Group A (r TMS group)
Device: Galvanic stimulation — galvanic stimulation of the vestibular apparatus
  Arms: Group B (Galvanic stimulation)

SUMMARY:
Vestibular disorders are disabling conditions that can have a major effect on functioning especially on daily activities and social participation. Latest epidemiological studies estimate that as many as 35% of adults aged 40 years or older had experienced some form of vestibular dysfunction. Non invasive brain stimulation techniques such as repetitive transcranial magnetic stimulation (rTMS) have been investigated as therapeutic interventions for various neurological disorders like motor deficits and balance disorders after various neurological deficits. The purpose of this study is to compare between rTMs stimulation and galvanic vestibular stimulation in patients with unilateral peripheral vestibular disorders.

DETAILED DESCRIPTION:
A pilot study has been recruited to calculate sample size and determine rTMs protocol that will be utilized during the study were two protocols has been compared and according to pilot study results collaborated with literature review a established protocol has been utilized. The subjects of both genders with age 30 to 60 will be allocated randomly into three equal groups A, B and C. Group A Outcomes measure will include : VNG (videonystagmography), Dizziness handicapped inventory, Berg balance scale, Vestibular disorders activities of daily living scale(VADL). Assessment will be done before and after treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis with unilateral peripheral vestibular disorders from audiologist or neurologist.
2. The patient's age will be ranged from thirty to sixty years old.
3. Patients will experience at least two symptoms of common symptoms of peripheral vestibular disorders.
4. Symptoms of vertigo and nystagmus lasting from seconds to one minute.
5. Vertigo that arises from changes in head position related to gravity.
6. Patients who experienced symptoms for more than three months (chronic patients)
7. Patients were selected to be ambulant.
8. Patients suffer from balance disturbance with low risk falling (41-56) and moderate risk falling ranges (21-40) according to berg balance scale.
9. All patients were medically stable, controlled with medical drugs for at least three months and failed to medical treatment with no other physical, mental or cognitive disorders.

Exclusion Criteria:

1. Benign positional vertigo.
2. Central vestibular disorders ( Ms, ataxia, migraine headache, posterior inferior cerebellar artery syndrome "PICA").
3. Vertigo that arises from changes in head position not related to gravity; as vertigo of cervical origin or vascular origin ( Vertebro- basilar insufficiency "VBI").
4. Previous surgery of the ear.
5. Bilateral peripheral vestibular weakness, central vestibular weakness, mixed vestibular weakness, or acute vestibular weakness.
6. Unstable health issues (cardiac dysfunction, end stage renal failure, unstable diabetes, uncontrolled hypertension >190/110…).
7. Pacemaker or other implanted electrically sensitive device.
8. Significant orthopedic or chronic pain syndrome (e.g any condition that wouldn't permit to completion of any of the tests).
9. Major cognitive dysfunction. neurodegenerative disease or major psychiatric condition ( Alzheimer's disease , depression….).
10. Chronic use of medications that could influence motor or sensory excitability (e.g AEDs, antipsychotic).
11. Alcohol abuse.
12. Epilepsy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Vestibular canal weakness | 1 mounth
  Videonystagmography- Scores ranging zero min score and 100 max score
Dizziness handicapped inventory | 1 month
  identify difficulties that you may be experiencing because of your dizziness- 25 items with max score 100 and min score zero

SECONDARY OUTCOMES:
Postural stability | 1 month
  Computerized dynamic Posturography- Scores ranging zero min score and 100 max score
Balance | 1 month
  Berg balance scale - 14 items each item scored from zero (min score)-4 (Max score) with total min score zero and max score 56
Vestibular disorders activities of daily living | 1 month
  The Vestibular Disorders Activities of Daily Living (VADL) scale assesses the impact of vestibular impairment on everyday activities. The 28 items are grouped into three dimensions: functional (self-care and intimate activities), ambulation (walking and stair climbing), and instrumental (home management and leisure activities).Each item is rated with zero (min score) to 10 (max score)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Giza Governorate, Egypt